CLINICAL TRIAL: NCT03902041
Title: The Prospective Randomized Controlled Clinical Study of Eltrombopag on Hematopoietic Reconstruction After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: The Prospective Randomized Controlled Study of Eltrombopag on Hematopoietic Reconstruction After Allogeneic HSCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Hematology Department, Shandong Provincial Hospital
Other Study IDs: SDPH001
Record Dates: First submitted 2019-03-30; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation; Eltrombopag
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment Group: The patients will receive Eltrombopag treatment after transplantation at d1.
  Interventions: Drug: Eltrombopag
- Control Group: The patients will not receive Eltrombopag treatment after transplantation.

INTERVENTIONS:
Drug: Eltrombopag — The patients will receive Eltrombopag treatment after transplantation
  Groups: Treatment Group

SUMMARY:
This study evaluates the addition of Eltrombopag after Hematopoietic stem cell transplantation (HSCT) to improve the engraftment of hematopoietic stem cell. Half of the participants will receive Eltrombopag,while the other will not receive the Eltrombopag.

DETAILED DESCRIPTION:
With the progress of transplantation technology，allogeneic hematopoietic stem cell transplantation is becoming an important treatment for hematological diseases and the long-term survival of patients is gradually improved. However, thrombocytopenia after transplantation has always been an important complication. Studies have shown that about 20% patients had different degrees of thrombocytopenia. Eltrombopag could promote hematopoietic stem cell proliferation and differentiation in vitro studies. It has also been widely used in the treatment of immune thrombocytopenia (ITP) and aplastic anemia(AA) and increased platelet levels in such diseases. Eltrombopag is also used to treat poor platelet engraftment after transplantation and the effective rate is about 60%-80%. Therefore, the application of Eltrombopag at early time after transplantation might promote platelet engraftment and reduce platelet transfusions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with definite diagnosis of hematological diseases, more than 30 kg, age18-60 years, gender and race are not limited;
2. Acceptance of allogeneic hematopoietic stem cell transplantation;
3. Voluntary acceptance of the study

Exclusion Criteria:

1. Patients with severe organ dysfunction or disease；
2. Patients who cannot tolerate oral Eltrombopag therapy;
3. Patients who refuse all-HSCT and Eltrombopag treatment;
4. Patients that investigator believed not suitable for enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients after allogeneic hematopoietic stem cell transplantation
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The engraftment of platelet | 3 years
  the day of platelet engraftment
The levels of platelet | 3 years
  The levels of platelet at 30 days after transplantation

SECONDARY OUTCOMES:
The number of platelet transfusions | 3 years
  The number of platelet units be transfused to the patients before platelet engraftment

OTHER OUTCOMES:
The engraftment of white blood cell | 3 years
  The day of white blood cell engraftment
OS | 3 years
  3years overall survival of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Heamtology Department, Provincial Hospital Affiliated to Shandong University, Jinan, Shandong, China